CLINICAL TRIAL: NCT00156169
Title: The Effect of the Alga Dunaliella Bardawil as a Source of 9-cis Retinoic Acid
Brief Title: The Effect of the Alga Dunaliella Bardawil as a Source of 9-cis Retinoic Acid on Lipid Profile in Fibrate Treated Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SHEBA-01-2358-AH-CTIL
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Low HDL Cholesterol
MeSH Terms: interventions — Cbr protein, Dunaliella

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dunaliella

SUMMARY:
The effect of fibrates on high density lipoprotein (HDL)-cholesterol levels is suggested to be mediated by its binding to peroxisome proliferator-activated receptor-g (PPARg). Upon ligand binding, PPARg heterodimerizes with the 9-cis retinoic acid receptor (RXR), and the heterodimer regulates gene expression. We assessed the hypothesis that a dual treatment with fibrate plus 9-cis b-carotene-rich powder of the alga Dunaliella bardawil, as a source of 9-cis retinoic acid, would improve the drug's effect on HDL-cholesterol levels.

patients with plasma HDL-cholesterol levels below 40 mg/dl and triglyceride (TG) levels above 200 mg/dl after fibrate treatment (for at least 6 weeks). are given four capsules of Dunaliella, providing 60 mg b-carotene/day. The all-trans to 9-cis b-carotene ratio in the capsules is about 1:1.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* Fibrate treatment (for at least 6 weeks)
* HDL-Cholesterol lower than 40mg/dl.
* Triglyceride over 150mg/dl.

Exclusion Criteria:

* High CPK.
* Elevated liver functions.
* Active CHD.
* Smokers.
* Diabetes patients treated with Insulin or Avandia. HbA1C great than 8.5.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-05; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Harari, Phd, Study Director — Sheba Medical Center